CLINICAL TRIAL: NCT06276478
Title: Positive Psychological Deconditioning of Pediatric Patients With Dental Anxiety Through Artificial Intelligence: Randomized Clinical Trial
Brief Title: Positive Psychological Deconditioning of Pediatric Patients With Dental Anxiety Through Artificial Intelligence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-PEDOAI
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Dental Anxiety; Dental Phobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental)
  Interventions: Other: AI-video
- Control group (Active Comparator)
  Interventions: Other: Verbal instructions

INTERVENTIONS:
Other: AI-video — Video administration for the explanation of the dental procedures followed by verbal instructions.
  Arms: Trial group
Other: Verbal instructions — Only verbal instructions will be administered for the explanation of the dental procedures
  Arms: Control group

SUMMARY:
Pediatric patients who will be attending dental treatment at both the Orthodontics and Pediatric Dentistry Unit, Department of Clinical, Surgical, Diagnostic, and Pediatric Sciences at the University of Pavia, Pavia, Italy and a private dental practice in Genoa, Italy, will be recruited for the study.

A cartoon version of a small molar will be drawn using the software Paint (version 22000.0, Microsoft Corporation, Redmond, Washington State, U.S.). The drawing will be animated using an AI-based software (Sketch MetaDemolab, Meta AI Research, Astor Place, New York city, New York, U.S.). A text will be created in collaboration with OpenAI (version 3.5, Open AI, San Francisco, California, U.S.) to be integrated into the video, utilizing terminology deemed most suitable for a patient with dental anxiety. The text will be transformed from written to spoken dialogue using an AI-based software (Flexclip, version 5.6.0, PearlMountain, Hong Kong, China), and then incorporated into the video.

Children will undergo the first dental visit at the baseline (T0), in which the following indexes will be assessed: Modified Dental Anxiety Scale (MDAS), Face-Leg-Activity-Cry-Consolability Scale (FLACC), Simplified Oral Hygiene Index (OHI-S), Bleeding on Probing (BOP) and the International Caries Detection and Assessment System (ICDAS). They will be randomly divided into two group:

* in the Trial group, patients will watch the the video, and then the tell-show-do technique will be used to explain the dental procedures;
* in the Control group, only the "tell-show-do" technique will be used. Variables considered will include age, gender, and the presence/absence of a parent or another companion.

At the second visit (T1), scheduled approximately after two weeks, the variables will be re-evaluated and professional debridement will be performed with a piezoelectric instrument (Satelect Acteon Newton p5 xs,Acteon Group, Mèrignac, France and Sonicflex Kavo, KaVo Dental, Biberach an der Riss, Germany) and manual scaler/curettes (Courette 9/10, 11/12 and 13/14 Gracey and Scaler lm 23, Hu Friedy, Europe). Values will be registered again, for the third time, after the professional debridement.

DETAILED DESCRIPTION:
The World Health Organization classifies dental phobia as a disease, making it a significant concern in the field of dentistry and a considerable challenge for practitioners. It has been included in the International Classification of Diseases (ICD-10) as one of the specific phobias. According to WHO estimates, it affects 15-20% of the population. Notably, it is estimated that over 50% of pediatric patients may exhibit varying degrees of anxiety during dental treatments. Therefore, it is desirable to develop methods to address this issue.

Existing literature already contains studies using anxiety control methods for pediatric patients. For example, in the review by S. L. Ainscough and colleagues, a study of 30 subjects aged 4 to 8 was cited, in which it was demonstrated that music can be an effective strategy to alleviate anxiety during dental sessions. In a previous study 13 subjects aged 11 to 16 were interviewed, showing how careful and optimal dentist-patient communication positively influences the approach to dental care. An illustrative study considered 150 randomly selected children aged 4 to 8, divided into five groups of 30 patients each. Anxiety was assessed using scales such as the Facial Image Scale and the Venham's Anxiety Scale, alongside physiological parameters like the physiological pulse rate. The study aimed to prove the effectiveness of modified tell-show-do techniques, such as tell-play-do, tell-play-do with a dentist smartphone game, tell-show-play-do, and ask-tell-ask.

Therefore, the objective of this study is to use Artificial Intelligence (AI) to provide a technique to positively decondition psychologically pediatric patients from the fear of dentists and make them more engaged and receptive to dental sessions with an animated cartoon created with AI with a dialogue tailored to pediatric patients with dental anxiety.

Pediatric patients who will be attending dental treatment at both the Orthodontics and Pediatric Dentistry Unit, Department of Clinical, Surgical, Diagnostic, and Pediatric Sciences at the University of Pavia, Pavia, Italy and a private dental practice in Genoa, Italy, will be recruited for the study.

A cartoon version of a small molar will be drawn using the software Paint (version 22000.0, Microsoft Corporation, Redmond, Washington State, U.S.). The drawing will be animated using an AI-based software (Sketch MetaDemolab, Meta AI Research, Astor Place, New York city, New York, U.S.). A text will be created in collaboration with OpenAI (version 3.5, Open AI, San Francisco, California, U.S.) to be integrated into the video, utilizing terminology deemed most suitable for a patient with dental anxiety. The text will be transformed from written to spoken dialogue using an AI-based software (Flexclip, version 5.6.0, PearlMountain, Hong Kong, China), and then incorporated into the video.

Children will undergo the first dental visit at the baseline (T0), in which the following indexes will be assessed: Modified Dental Anxiety Scale (MDAS), Face-Leg-Activity-Cry-Consolability Scale (FLACC), Simplified Oral Hygiene Index (OHI-S), Bleeding on Probing (BOP) and the International Caries Detection and Assessment System (ICDAS). They will be randomly divided into two group:

* in the Trial group, patients will watch the the video, and then the tell-show-do technique will be used to explain the dental procedures;
* in the Control group, only the "tell-show-do" technique will be used. Variables considered will include age, gender, and the presence/absence of a parent or another companion.

At the second visit (T1), scheduled approximately after two weeks, the variables will be re-evaluated and professional debridement will be performed with a piezoelectric instrument (Satelect Acteon Newton p5 xs,Acteon Group, Mèrignac, France and Sonicflex Kavo, KaVo Dental, Biberach an der Riss, Germany) and manual scaler/curettes (Courette 9/10, 11/12 and 13/14 Gracey and Scaler lm 23, Hu Friedy, Europe). Values will be registered again, for the third time, after the professional debridement.

ELIGIBILITY:
Inclusion Criteria:

* age between 5 and 10 years
* Modified Dental Anxiety Scale (MDAS) (Humphris GM et al. 1995) greater than or equal to children must score equal to or higher than 19 in the questionnaire based on the "The modified dental anxiety scale."
* FLACC score (Merkel, S. I. et al., 1997) greater than or equal to 4
* Simplified Oral Hygiene Index (OHI-S) (Greene JC et al, 1964) greater than or equal to 1.3.

Exclusion Criteria:

* Previous Traumatic Dental/Orthodontic Treatments
* Previous Hospitalizations
* Intellectual Disabilities and Psychiatric Disorders

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Change in Modified Dental Anxiety Scale - MDAS (Humphris GM et al. 1995) | Baseline (T0) and after 14 days (T1)

SECONDARY OUTCOMES:
Change in Face, Leg, Activity, Cry, Consolability Scale - FLACC (Merkel, S. I. et al., 1997) | Baseline (T0) and after 14 days (T1)
Change in Bleeding on Probing - BoP (Löe H. et al.,1967) | Baseline (T0) and after 14 days (T1)
Change in Simplified Oral Hygiene Index - OHI-S (Greene JC et al, 1964) | Baseline (T0) and after 14 days (T1)
International Caries Detection and Assessment System - ICDAS | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, MSc, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.